CLINICAL TRIAL: NCT04345354
Title: Observational Study of the Value of Using Continuous Positive Airway Pressure (CPAP) Ventilation on the Occurrence of Respiratory and Cardiovascular Complications in Patients at High Risk of Obstructive Apnea Syndrome During Postoperative Sleep Surgery of a Major Abdominal Surgery.
Brief Title: Observational Study of the Value of Using Obstructive Sleep Apnea-hypopnea Syndrome (CPAP) Ventilation on the Occurrence of Respiratory and Cardiovascular Complications in Patients at High Risk of Obstructive Apnea Syndrome During Postoperative Sleep Surgery of a Major Abdominal Surgery.
Acronym: APNOSIS-BIS
Status: Completed | Type: Observational
Sponsor: Poitiers University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: APNOSIS-BIS
Record Dates: First submitted 2018-08-06; First posted 2020-04-14 (Actual); Last update posted 2020-04-14 (Actual); Status verified 2020-04

CONDITIONS: Major Abdominal Surgery

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patient with continuous positive airway pressure treatment
- without continuous positive airway pressure treatment

SUMMARY:
The presence of an obstructive sleep apnea-hypopnea syndrome (OSAHS) is a perfectly identified cardiovascular and metabolic risk factor responsible for excess mortality in patients with severe OSAHS, while life expectancy, when the SAHOS is treated by continuous positive airway pressure (CPAP) is close to that of the general population. It also represents a factor of excess mortality, little known and poorly explored, in relation to morbidity and mortality occurring during the perioperative period accompanying any general anesthesia.

ELIGIBILITY:
Inclusion Criteria:

* Patients over 18 years old and naive to any treatment with obstructive sleep apnea-hypopnea syndrome,
* Patients at high risk of obstructive sleep apnea-hypopnea syndrome (STOP BANG ≥ 3),
* Patients scheduled for major abdominal surgery (all intraperitoneal surgeries excluding vesicles, eventrations and hernias, all aortic surgeries excluding endovascular surgeries) within a minimum of 10 days,
* It is possible to integrate the explanations concerning the realization of the ApneaLink ™ Air in autonomy and to ensure its restitution under 24-48h,

Exclusion Criteria:

* Patients with obstructive sleep apnea-hypopnea syndrome diagnosed before surgery,
* Patients with heart failure (NYHA> II),
* Patients with moderate to severe COPD
* Patients participating in a clinical trial,

Ages: 18 Years to 100 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients without known obstructive sleep apnea-hypopnea syndrome, presenting at anesthesia consultation for visceral surgery to be performed at least within 10 days.
Sampling Method: Probability Sample
Enrollment: 48 (Actual)
Dates: Start 2016-06-14 (Actual); Primary Completion 2018-12 (Actual); Study Completion 2018-12 (Actual)

PRIMARY OUTCOMES:
Evaluate rate of respiratory complications with moderate sleep apnea syndrome with continuous positive airway pressure treatment | 7 days
Evaluate rate of respiratory complications with moderate sleep apnea syndrome without continuous positive airway pressure treatment | 7 days
Evaluate rate of cardiovascular complications with moderate sleep apnea syndrome with continuous positive airway pressure treatment | 7 days
Evaluate rate of cardiovascular complications with moderate sleep apnea syndrome without continuous positive airway pressure treatment | 7 days

SECONDARY OUTCOMES:
Evaluate tolerance and observance of continuous positive airway pressure treatment | 7 days
Evaluate the feasibility of the ApneaLink | 7 days
Evaluate the prevalence of obstructive sleep apnea-hypopnea syndrome patients to the severity level of the STOPBANG score, | 7 days
Evaluate the duration and place of hospitalization during the post-surgical course | 28 days

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Claude MEURICE, Principal Investigator — Poitiers University Hospital
Locations (1):
- Chu de Poitiers, Poitiers, France

IPD SHARING:
Plan to Share IPD: No